CLINICAL TRIAL: NCT02809235
Title: The Role of Cholecystokinin and the Cholecystokinin Receptor in the Airway Smooth Muscle of Asthmatics
Brief Title: Fatty Acids in Airway Smooth Muscle of Asthmatics
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Elliot Israel, MD, Elliot Israel, MD, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016P000273
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2024-10-23 (Actual); Status verified 2023-11

CONDITIONS: Asthma
Keywords: asthma; smooth muscle; lauric acid; dietary supplement
MeSH Terms: conditions — Asthma | interventions — Coconut Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- coconut oil (Experimental): Subjects will be instructed to supplement their diet with 3 tablespoons of coconut oil daily for three weeks.
  Interventions: Dietary Supplement: coconut oil

INTERVENTIONS:
Dietary Supplement: coconut oil — 3 tablespoons per day of supplemental coconut oil

SUMMARY:
In this proof of concept study, the investigators aim to determine if supplementation with coconut oil causes an increase in cholecystokinin and cholecystokinin receptor expression in the airway smooth muscle of lean asthmatics, and whether these changes correlate with changes in airway stiffness (estimated by bronchodilator reversibility, airway reactivity, and airway resistance) or symptom control.

The investigators propose a 5 week, single center trial in 20 lean patients with mild asthma (not taking inhaled corticosteroids) aged 18 and older. Subjects will supplement their usual diets with 3 tablespoons of coconut oil, a commercially available oil with high dodecanoic acid content, for 3 weeks. To quantify changes in airway smooth muscle cholecystokinin and cholecystokinin-receptor expression, each subject will undergo bronchoscopy with endobronchial biopsies before and after coconut oil ingestion.

For the secondary analysis, subjects will also complete spirometry with bronchodilator testing, methacholine challenge, body plethysmography, and an Asthma Control Questionnaire (ACQ) before and after the dietary intervention. This information will be used to compare the changes in airway smooth muscle cholecystokinin and cholecystokinin receptor expression to changes in bronchodilator reversibility, airway reactivity, airway resistance, and symptom control.

In the exploratory aims, the investigators will correlate the changes in airway smooth muscle cholecystokinin and cholecystokinin receptor expression with changes in FEV1 and peak flow measurements.

The investigators therefore hope to elucidate information about the mechanistic role of cholecystokinin in airway smooth muscle stiffness and contraction.

DETAILED DESCRIPTION:
20 lean (BMI<25) nonsmokers at least 18 years of age with mild asthma will be recruited from the Asthma Research Center database. A sample size of 12 asthmatics is needed to have 80% power to detect a 3-fold increase in cholecystokinin (CCK) post dodecanoic acid ingestion at alpha level of 0.05, assuming the standard deviation is ≤2.25 in cycle scale. To account for probable incomplete retention, 20 subjects will be recruited. While the calculated standard deviation is 1.775, the investigators chose to base our calculations off of a larger standard deviation because of our small sample size.

Study subjects will be asked to come to 5 visits, described in detail below.

Visit 1: Eligibility Screen Pre-screened Volunteers will be asked not to take their short acting bronchodilators or ipratropium within 6 hours of this visit. They will complete a medical history that includes detailed information about past and current asthma medications, ACQ, physical exam with weight/BMI check and spirometry with bronchodilator testing. They will undergo body plethysmography to measure baseline airway resistance.

Visit 2: Eligibility Screen, methacholine challenge Subjects will return at any point during the 1-4 weeks allowed between visits 1 and 3. They will be told to not to take their short acting bronchodilators or ipratropium within 8 hours of this visit and to avoid caffeine (coffee, tea, cola drinks, and chocolate) the day of the visit. This visit will be short, comprised only of a methacholine challenge, to measure baseline airway reactivity.

Visit 3: Bronchoscopy Eligible subjects will be asked not to take aspirin, anticoagulant (e.g., warfarin) or antiplatelet (e.g., clopidogrel) medication in the 7 days prior to this second visit. They will also be told not to eat or drink within 6hrs of the visit.

At the beginning of the visit, subjects will be instructed on how to use a peak flow meter. Baseline peak flow measurements will be recorded. They will then undergo bronchoscopy with endobronchial biopsy. The investigators will perform laser capture on the biopsy samples to isolate the smooth muscle cells and quantify the cells' CCK and cholecystokinin receptor (CCK-AR) content via quantitative polymerase chain reaction (PCR).

The study participants will then be instructed to supplement their usual diets with 3 tablespoons of coconut oil (about 21.6g dodecanoic acid, 375 calories) daily for three weeks. The oil should be consumed uncooked so that its chemical form is unaltered. It can be swallowed by tablespoon or mixed into/spread on foods. The investigators recommend that it take the place of other fatty foods rather than be added to each subject's diet, so that subjects' overall daily caloric intake does not increase (and so that subjects do not gain weight).

The average adult ingests 0.8g of dodecanoic acid daily, according to a 2004 NHANES report. Dodecanoic acid is present at particularly high concentration in coconut oil (50% dodecanoic acid by weight). While the degree to which ingested dodecanoic acid reaches plasma and airway smooth muscle cells is unknown, prior trials confirm rise in plasma concentration of similar fatty acids (including gama linolenic acid, stearidonic acid, alpha linolenic acid, and eicosapentaenoic acid) after supplementation with as little as 0.25-4g daily for 3 weeks. The investigators have chosen to maximize the supplemented dose (to about 20g) so that any possible effect of dodecanoic acid on the airway smooth muscle is not missed. The 3 week duration is modeled after the aforementioned studies.

The investigators will provide each subject with a Drug Diary and peak flow meter. Subjects will be instructed to keep track of their daily coconut oil ingestion and peak flow measurements. They will be told to measure peak flow daily between 5 and 11 am, prior to the use of any morning inhalers, and to call the study coordinators if they experience a change in their asthma symptoms or if their measurements drop by more than 20% of their baseline. In addition, a study investigator will call each subject weekly to encourage compliance and to ensure that the subject has no questions or adverse events.

Visit 4: Followup exam, ACQ, pulmonary function tests After 3 weeks of coconut oil ingestion, subjects will return for a repeat physical exam with weight/BMI check and methacholine challenge. They will fill out a second ACQ and continue to supplement their diet with coconut oil until visit 5.

Visit 5: Followup pulmonary function tests, second bronchoscopy Subjects will return 1-3 days later for visit 5. They will again be told not to take aspirin, anticoagulant (e.g., warfarin) or antiplatelet (e.g., clopidogrel) medication in the 7 days prior to this final visit, and not to eat or drink within 6hrs of the visit.

The investigators will formally review each subject's Drug Diary and peak flow measurements. Eligible subjects will undergo spirometry, bronchodilator reversibility testing, body plethysmography, and bronchoscopy with endobronchial biopsy. The investigators will process the samples and compare the post-fatty acid ingestion outcomes to the baseline values.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants, age 18 years and older at enrollment
2. Never smokers or <10 pack year smoking history
3. Body mass index (BMI) <25
4. Clinical history consistent with asthma for >1 year
5. No use of an inhaled corticosteroid in the prior 3mo
6. Ability to perform reproducible spirometry according to ATS criteria
7. Baseline Forced expiratory volume in 1 second (FEV1) ≥ 60% predicted
8. Presence of bronchodilator reversibility, as defined by a minimum of 12% and ≥ 200 ml improvement after 4 puffs of albuterol, each 90 μg
9. Ability to provide informed consent, as evidenced by signing a copy of the consent form approved by the Institutional Review Board.

Exclusion Criteria:

1. Supplementation with fatty acids within the last 3 months
2. BMI ≥25
3. Pregnant or nursing
4. History of smoking (cigarettes, cigars, pipes, marijuana or any other substances) within the past 1 year, or >10 pack-years total
5. Use of inhaled corticosteroid in the prior 3 mo
6. Lack of bronchodilator response to 4 puffs of albuterol
7. Medical contraindication to bronchoscopy/biopsy, i.e inability to stop aspirin, anticoagulant, or antiplatelet at any point during the study; coagulopathy; inability to lay flat; asthma exacerbation requiring corticosteroids in the preceding 4 weeks; history of adverse reaction or allergy to sedatives; history of difficult airway, or past difficulty with intubation
8. Major medical problems prohibiting study participation, i.e presence of chronic or active lung disease other than asthma or history of unstable significant medical illness other than asthma
9. Evidence that the participant may be non-adherent to medication regimen, or may move from the performance site area before trial completion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-11 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Change in Airway Smooth Muscle (ASM) Cholecystokinin (CCK) and Cholecystokinin Receptor (CCK-AR) expression with coconut oil supplementation | 3 weeks

SECONDARY OUTCOMES:
Change in ASM CCK and CCK-AR expression with coconut oil supplementation, versus change in bronchodilator reversibility. | 3 weeks
Change in ASM CCK and CCK-AR expression with coconut oil supplementation, versus change in bronchial hyperresponsiveness (PC20). | 3 weeks
Change in ASM CCK and CCK-AR expression with coconut oil supplementation, versus change in airway resistance | 3 weeks
Change in ASM CCK and CCK-AR expression with coconut oil supplementation, versus change in Asthma Control Questionnaire (ACQ) score. | 3 weeks

OTHER OUTCOMES:
Change in ASM CCK and CCK-AR expression with coconut oil supplementation, versus change in Forced Expiratory Volume in 1 second (FEV1). | 3 weeks
Change in ASM CCK and CCK-AR expression with coconut oil supplementation, versus change in peak flow. | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Israel, MD, Principal Investigator — Asthma Research Center
Locations (1):
- Asthma Research Center, Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided